CLINICAL TRIAL: NCT04999020
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Ravulizumab in Adult Participants With Dermatomyositis
Brief Title: Ravulizumab Versus Placebo in Adult Participants With Dermatomyositis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1210-DM-310; 2021-001200-15 (EudraCT Number)
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Dermatomyositis
Keywords: Ravulizumab; ALXN1210; Ultomiris; Pharmacokinetics; Pharmacodynamics; Efficacy; DM
MeSH Terms: conditions — Dermatomyositis | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): Participants will receive ravulizumab in both Parts A and B.
  Interventions: Drug: Ravulizumab
- Placebo (Placebo Comparator): Participants will receive placebo in both Parts A and B.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravulizumab — Intravenous dosing will consist of a loading dose followed by maintenance doses administered every 8 weeks (q8w). The maintenance dosing will be initiated 2 weeks after the loading dose is administered.
  Other Names: ALXN1210; Ultomiris
  Arms: Ravulizumab
Drug: Placebo — Intravenous dosing will consist of a loading dose followed by maintenance doses administered q8w. The maintenance dosing will be initiated 2 weeks after the loading dose is administered.
  Arms: Placebo

SUMMARY:
This is a Phase 2/3, double-blind, randomized, placebo-controlled, parallel group, multicenter study to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of ravulizumab in adult participants with dermatomyositis (DM).

DETAILED DESCRIPTION:
The study will be conducted in 2 parts: Part A (Phase 2) and Part B (Phase 3). There will be 3 periods in both Part A and Part B of this study: Screening Period, Randomized Controlled Period, and Open-Label Extension Period.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older at the time of signing the informed consent.
* Body weight ≥ 30 kilograms at the time of Screening.
* Male or female.
* Diagnosis: Meet 2017 American College of Rheumatology/European League Against Rheumatism classification criteria for definite or probable DM.
* Participants who have an inadequate response or are intolerant to 1 or more DM treatments, including systemic corticosteroids or immunosuppressive/immunomodulatory therapies (for example, azathioprine, methotrexate, rituximab, intravenous immunoglobulin), either in combination or as monotherapy.
* Vaccinated against Neisseria meningitidis within 3 years prior to initiating ravulizumab as per national and local guidelines. Participants must receive the vaccination at least 2 weeks before first study intervention. The sponsor recommends that national and local guidelines for prophylactic antibiotics should also be followed.
* Female participants of childbearing potential and male participants must follow specified contraception guidance as described in the protocol.

Key Exclusion Criteria:

* Participants who have been diagnosed with cancer within the last 3 years need to have appropriate negative cancer screening as per local standard of care within 6 months before Screening (basal or squamous cell skin cancer or carcinoma in situ of the cervix needs to have been excised and without evidence of residual disease for at least 3 months before Screening).
* Evidence of active malignant disease or malignancies diagnosed within the previous 3 years including hematological malignancies and solid tumors.
* Participants with other forms of myositis.
* As per investigator discretion, participants with significant muscle damage (for example, severe muscle atrophy, end stage muscle disease, MRI with severe atrophy or fibrofatty replacement)
* History of Neisseria meningitidis infection.
* Human immunodeficiency virus (HIV) infection (evidenced by HIV Type 1 or Type 2 antibody titer).
* Active systemic bacterial, viral, or fungal infection within 14 days prior to ravulizumab administration.
* Presence of fever ≥ 38°Celsius (100.4°Fahrenheit) within 7 days prior to study drug administration on Day 1.
* History of hypersensitivity to murine proteins or to 1 of the excipients of ravulizumab.
* Pregnant, breastfeeding, or intending to conceive during the course of the study.
* Inability or unwillingness to adhere to the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (100):
- United States (20):
  - Research Site, Phoenix, Arizona
  - Research Site, Irvine, California
  - Research Site, Santa Monica, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Fairway, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Las Vegas, Nevada
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, North Richland Hills, Texas
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Camperdown
  - Research Site, Murdoch
- Brazil (11):
  - Research Site, Belém
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Juiz de Fora
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Serra
  - Research Site, Vitória
- France (6):
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (7):
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Jena
- Italy (18):
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Iesi
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Rozzano
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Torrette AN
  - Research Site, Udine
  - Research Site, Verona
- Japan (10):
  - Research Site, Bunkyō City
  - Research Site, Hiroshima
  - Research Site, Iruma-Gun
  - Research Site, Nagoya
  - Research Site, Narita-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Urayasu-shi
- Research Site, Warsaw, Poland
- South Korea (3):
  - Research Site, Daejeon
  - Research Site, Junggu
  - Research Site, Seoul
- Spain (12):
  - Research Site, A Coruña
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taoyuan
- Turkey (Türkiye) (2):
  - Research Site, Altındağ-Ankara
  - Research Site, Istanbul
- United Kingdom (5):
  - Research Site, Edinburgh
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Salford
  - Research Site, West Bromwich

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-DM-310&attachmentIdentifier=e7eaf251-b584-4aa0-825a-6753743274b8&fileName=ALXN1210-DM-310_Abbreviated_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts - Part A and Part B. The study was terminated early and participants were not enrolled into Part B. Therefore, results are presented for Part A of the study only. Part A consisted of a Randomized Controlled Period (RCP) and an Open-Label Extension (OLE) period.
Groups:
- RCP: Ravulizumab: Participants received a loading dose of ravulizumab on Day 1 followed by a maintenance dose at Week 2 and then ravulizumab once every 8 weeks (Q8W) during the 26-week RCP.
- RCP: Placebo: Participants received placebo on Day 1, and Weeks 2, 10, and 18 during the 26-week RCP.
- OLE: Ravulizumab to Ravulizumab: Participants who received ravulizumab during the RCP continued to receive ravulizumab during the 130-week OLE. Participants received a blinded ravulizumab dose at Week 26, a maintenance dose at Week 28, then ravulizumab Q8W for the remainder of the OLE period.
- OLE: Placebo to Ravulizumab: Participants who received placebo during the RCP received ravulizumab during the 130-week OLE. Participants received a blinded ravulizumab dose at Week 26, a maintenance dose at Week 28, then ravulizumab Q8W for the remainder of the OLE period.
Period: Randomized Controlled Period (RCP)
Arm/Group | RCP: Ravulizumab | RCP: Placebo | OLE: Ravulizumab to Ravulizumab | OLE: Placebo to Ravulizumab
Started | 26 | 12 | 0 (Data is presented in this period for the participants in the RCP only.) | 0 (Data is presented in this period for the participants in the RCP only.)
Received at Least 1 Dose of Treatment | 26 | 12 | 0 (Data is presented in this period for the participants in the RCP only.) | 0 (Data is presented in this period for the participants in the RCP only.)
Completed | 22 | 9 | 0 (Data is presented in this period for the participants in the RCP only.) | 0 (Data is presented in this period for the participants in the RCP only.)
Not Completed | 4 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Period: Open-Label Extension (OLE) Period
Arm/Group | RCP: Ravulizumab | RCP: Placebo | OLE: Ravulizumab to Ravulizumab | OLE: Placebo to Ravulizumab
Started | 0 (Data is presented in this period for the participants in the OLE only.) | 0 (Data is presented in this period for the participants in the OLE only.) | 22 | 9
Received at Least 1 Dose of Treatment | 0 (Data is presented in this period for the participants in the OLE only.) | 0 (Data is presented in this period for the participants in the OLE only.) | 22 | 9
Completed | 0 (Data is presented in this period for the participants in the OLE only.) | 0 (Data is presented in this period for the participants in the OLE only.) | 0 | 0
Not Completed | 0 | 0 | 22 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 17 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Groups:
- Ravulizumab: Participants received a loading dose of ravulizumab on Day 1 followed by a maintenance dose at Week 2 and then Q8W during the 26-week RCP.
- Placebo: Participants received placebo on Day 1, Weeks 2, 10 and 18 during the 26-week RCP.
- Total: Total of all reporting groups
Arm/Group | Ravulizumab | Placebo | Total
Number analyzed (Participants) | 26 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.38) | 59.3 (9.31) | 53.4 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 27
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 23 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 10 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With International Myositis Assessment and Clinical Studies Total Improvement Score (IMACS-TIS) (TIS40) Response at Week 26 of the Randomized Controlled Period
Description: Data are presented for the number of participants with a TIS40 response, defined as an IMACS-TIS score ≥ 40 at Week 26. IMACS-TIS is a clinical instrument that encompasses 6 core set measure (CSMs) (physician, patient, extra-muscular global activity, muscle strength, Health Assessment Questionnaire [HAQ], and muscle enzyme levels). A Total Improvement Score (TIS: 0-100), was determined by summing scores in each CSM, and was based on the improvement and relative weight of each CSM. A higher score indicated greater improvement. TIS40 was considered a moderate improvement score.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 9 | 6
Statistical Analysis 1: Comparison: RCP: Ravulizumab vs RCP: Placebo; Test type: Superiority; p = 0.4192, Barnard's unconditional exact test; Difference in response rates = -15.38, 80% CI 2-sided [-38.55 to 8.48]

2. Secondary Outcome: TIS at Week 26
Description: TIS scores ranged from 0-100 with higher scores indicating a greater improvement. Scores were determined by summing scores in each of the 6 CSMs of the IMAC (physician, patient, extra-muscular global activity, muscle strength, HAQ, and muscle enzyme levels). Clinically meaningful thresholds for improvement were defined as ≥ 20 point improvement response on IMACS-TIS (TIS20; mild), ≥ 40 point improvement response on IMACS TIS (TIS40; moderate) and ≥ 60 point improvement response on IMACS-TIS (TIS60; severe). Scores were based on the improvement and relative weight of each CSM. Data are presented for TIS (least squares mean) at Week 26.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group. Overall number of participants analyzed = participants with evaluable data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | 31.16 (4.185) | 43.28 (6.650)

3. Secondary Outcome: Change From Baseline In Cutaneous Dermatomyositis Disease Area And Severity Index (CDASI) Activity Score at Week 26
Description: The CDASI is an instrument that separately measures activity and damage in the skin of dermatomyositis (DM) participants. It contains 3 activity measures (erythema, scale, and erosion/ulceration) and 2 damage measures (poikiloderma and calcinosis). CDASI score is calculated by rating the severity of skin disease in 15 anatomical locations on the body based on the activity and damage components. CDASI was completed by the Clinician or Clinician-Investigator while examining the participant. Total CDASI scores ranged from 0-100, with higher scores indicating a greater disease severity. Change from baseline in CDASI Total Activity Score at Week 26 was analyzed using a mixed model repeated measures (MMRM). The MMRM model included the observed Total Activity Score values at post baseline visits (Week 26) as the dependent variable.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | -3.80 (1.249) | -7.47 (2.021)

4. Secondary Outcome: Number of Participants With Response Related to Muscle Enzymes: Normalization of Most Abnormal Baseline Enzyme at Week 26
Description: Laboratory tests were conducted to measure serum activities of muscle associated enzymes including creatine kinase (CK), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactate dehydrogenase (LDH), and aldolase. Data are presented for the number of participants who had an abnormal muscle enzyme at baseline that had been normalized at Week 26.
Time Frame: Baseline, Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 4 | 1

5. Secondary Outcome: Change From Baseline In IMACS CSMs: Extra-Muscular Disease Activity Based on Myositis Disease Activity Assessment Tool (MDAAT) at Week 26
Description: The MDAAT assesses disease activity of extra-muscular organ systems and muscles in participants with DM. The validated MDAAT tool measures the degree of disease activity of extra-muscular organ systems and muscle on a 0-10 centimeter (cm) visual analog scale (VAS). Extra-muscular activity ranged between 0 and 10, where, 0 cm = absent and 10 cm = maximum disease activity.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | -0.92 (0.383) | -2.13 (0.614)

6. Secondary Outcome: Change From Baseline In IMACS CSMs: Physician Global Activity Assessment at Week 26
Description: The physician global activity assessment provides an overall rating of disease activity related to myositis. Disease activity is judged by the physician based on all information available at the time of evaluation, including the participant's appearance, medical history, physical examination, laboratory testing, and prescribed medical therapy. The global disease activity score is recorded on a 10-cm VAS, where 0 cm= no evidence of disease activity and 10 cm= extremely severe disease activity.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | -1.18 (0.413) | -1.97 (0.649)

7. Secondary Outcome: Change From Baseline In IMACS CSMs: Patient Global Activity Assessment at Week 26
Description: The patient global activity assessment provides an overall rating of disease activity related to myositis from the participant's perspective. Participants were asked to consider all of the active inflammation in their own muscles, skin, joints, intestines, heart, lungs, or other parts of the body that can improve with treatment. The patient global disease activity score was recorded on a 10-cm VAS that contained a smiley face at the 0-cm anchor and a sad face at the 10 cm anchor to help participants understand the scale. Scores ranged from 0 (no evidence of disease activity) to 10 (extremely active or severe disease activity).
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | -1.43 (0.432) | -1.12 (0.699)

8. Secondary Outcome: Change From Baseline In IMACS CSMs: Manual Muscle Testing Subset 8 Muscles (MMT-8) at Week 26
Description: The purpose of the MMT-8 was to measure muscle strength as part of the physical examination. It included a subset of 8 muscle groups: neck flexors, deltoids, biceps, wrist, extensors, gluteus maximus and medius, quadriceps, and ankle dorsiflexors. Total MMT8 scores ranged from 0 (lowest strength) to 150 (highest strength).
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | 9.5 (1.85) | 12.6 (2.98)

9. Secondary Outcome: Change From Baseline In IMACS CSMs: Health Assessment Questionnaire (HAQ) at Week 26
Description: The HAQ is a brief self-report questionnaire that assesses physical function pertaining to activities of daily living in a variety of domains. The HAQ includes 20 questions relating to 8 domains of function: dressing and grooming, arising, eating, walking, hygiene, reach, grip and usual activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific subcategory items. The standard disability score is calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do), with higher values indicating higher disability.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 25 | 12
scores on a scale | -0.1289 (0.08607) | -0.4188 (0.13676)

10. Secondary Outcome: Number of Participants With CDASI Response (>=7-point Improvement) at Week 26
Description: The CDASI is an instrument that separately measures activity and damage in the skin of dermatomyositis (DM) participants. It contains 3 activity measures (erythema, scale, and erosion/ulceration) and 2 damage measures (poikiloderma and calcinosis). CDASI score is calculated by rating the severity of skin disease in 15 anatomical locations on the body based on the activity and damage components. CDASI was completed by the Clinician or Clinician-Investigator while examining the participant. Total CDASI scores ranged from 0-100, with higher scores indicating a greater disease severity.
  Data are presented for the number of participants with a CDASI response. Response was defined as a >=7 point improvement in participants who did not have an intercurrent event at or prior to the relevant timepoint.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 6 | 4

11. Secondary Outcome: Number of Participants With Cutaneous Dermatomyositis Activity Physician's Global Assessment (CDA-IGA) Response at Week 26
Description: CDA-IGA is a scale that was created to measure disease severity in participants with skin disease. It is a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) with morphologic descriptors for each score. The CDA-IGA was completed by the Investigator and was used to describe the overall appearance of lesions at a given time point. Data are presented for the number of participants with a CDA-IGA response at Week 26. A response was defined as participants with clear or almost clear skin (score of 0 or 1) who did not have an intercurrent event at or before the relevant timepoint.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 5 | 2

12. Secondary Outcome: Number of Participants With ≥ 20-Point Improvement Response on IMACS-TIS (TIS20) Response at Week 26
Description: TIS20 was defined as a ≥20-point improvement response on IMACS-TIS. IMACS-TIS is a clinical instrument that encompasses 6 CSMs (physician, patient, extra-muscular global activity, muscle strength, HAQ, and muscle enzyme levels). A Total Improvement Score (TIS: 0-100), was determined by summing scores in each CSM, and was based on the improvement and relative weight of each CSM. Higher scores indicated greater improvement/response. TIS20 is considered a mild improvement score.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 14 | 9

13. Secondary Outcome: Number of Participants With ≥ 60-Point Improvement Response on IMACS-TIS (TIS60) Response at Week 26
Description: TIS60 was defined as a ≥60-point improvement response on IMACS-TIS. IMACS-TIS is a clinical instrument that encompasses 6 CSMs (physician, patient, extra-muscular global activity, muscle strength, HAQ, and muscle enzyme levels). A Total Improvement Score (TIS: 0-100), was determined by summing scores in each CSM, and was based on the improvement and relative weight of each CSM. Higher scores indicated greater improvement/response. TIS60 is considered a severe improvement score.
Time Frame: Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 3 | 2

14. Secondary Outcome: Time to First Response of TIS20, TIS40, or TIS60
Description: TIS20, 40 and 60 were defined as a ≥20, ≥40 and ≥60-point improvement response on IMACS-TIS respectively. IMACS-TIS is a clinical instrument that encompasses 6 CSMs (physician, patient, and extra-muscular global activity, muscle strength, HAQ, and muscle enzyme levels). A Total Improvement Score (TIS: 0-100), was determined by summing scores in each CSM, and was based on the improvement and relative weight of each CSM. Higher scores indicated greater improvement/response. TIS20, 40 and 60 were considered mild, moderate and severe improvement scores respectively. Data are presented for the time to first response of TIS20, TIS40, or TIS60. The median time to TIS20, TIS40, and TIS60 was defined at the time in which 50% of the participants experienced TIS20, TIS40, or TIS60, respectively, based on a Kaplan-Meier analysis.
Time Frame: Baseline through Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group. Overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participant evaluable for the specified category.
Measure: Median (80% Confidence Interval); unit: weeks
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
weeks
  Time to TIS20 | 10.43 [10.14 to 17.86] | 10.14 [2.14 to 10.14]
  Time to TIS40 | 25.86 [18.14 to NA] — As fewer than 50% of the participants experienced the event of TIS40 and the median time to TIS40 event was close to the maximum follow-up period, there was not enough information on longer follow-up times to estimate the upper bound of the confidence interval. | 26.0 [10.14 to 26.29]
  Time to TIS60 | NA [NA to NA] — As fewer than 50% of the participants in the arm experienced TIS60 response during the RCP (the Week 26 period), the median time could not be estimated along with the associated 80% confidence intervals using Kaplan-Meier analysis. | NA [26.14 to NA] — As fewer than 50% of the participants in the arm experienced TIS60 response during the RCP (the Week 26 period), the median time could not be estimated along with the associated upper 80% confidence interval using Kaplan-Meier analysis.

15. Secondary Outcome: Number of Participants With Clinical Worsening (CW) During the RCP At 2 Consecutive Visits
Description: CW was defined as one of the following:
  1. Physician's global activity VAS worsening ≥ 2 cm and MMT-8 worsening ≥ 20% compared to baseline
  2. Global extra muscular activity worsening ≥ 2 cm on the MDAAT VAS compared to baseline
  3. Any 3 of 5 CSMs (excluding muscle enzymes) worsening by ≥ 30% compared to baseline
  Data are presented for the number of participants with clinical worsening during the RCP at 2 consecutive visits.
Time Frame: Baseline through Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 2 | 0

16. Secondary Outcome: Number of Participants Who Received Acute Rescue Therapy With Standard DM Treatment
Description: Acute rescue therapy with standard DM treatment included an increased dose of a medication that was being taken for DM or the initiation of a new DM treatment (glucocorticoid and/or immunosuppressive/immunomodulatory therapy [ISTs]). Data are presented for the number of participants who received acute rescue therapy with standard DM treatment.
Time Frame: Baseline through Week 26
Population: Randomized Set, which included all randomized participants grouped by randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | RCP: Ravulizumab | RCP: Placebo
Number analyzed (Participants) | 26 | 12
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 130 weeks
Description: Safety Set for the RCP, which included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention received. One participant who was randomized to ravulizumab during the RCP received placebo. This participant was analyzed in the placebo group for safety data collection and reporting.
  OLE Set for the OLE period, which included all randomized participants who received at least 1 dose of ravulizumab from Week 26 onward.
Arm/Group | RCP: Ravulizumab | RCP: Placebo | OLE: Ravulizumab to Ravulizumab | OLE: Placebo to Ravulizumab
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/13 | 0/22 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/13 | 4/22 | 4/9
Other Adverse Events (participants affected / at risk) | 9/25 | 10/13 | 11/22 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RCP: Ravulizumab (N=25) | RCP: Placebo (N=13) | OLE: Ravulizumab to Ravulizumab (N=22) | OLE: Placebo to Ravulizumab (N=9)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/18 | 0/9 | 1/16 | 0/6 — Number at risk has been adjusted as this is a sex-specific event.
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RCP: Ravulizumab (N=25) | RCP: Placebo (N=13) | OLE: Ravulizumab to Ravulizumab (N=22) | OLE: Placebo to Ravulizumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tongue movement disturbance (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Vaccination site swelling (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1
COVID-19 (Infections and infestations) | 2 | 3 | 2 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Pyoderma (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 2 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Part A did not meet its primary endpoint and the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04999020/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT04999020/SAP_001.pdf